CLINICAL TRIAL: NCT02268721
Title: Food'to'Go - a Feasibility Study of Post-discharge Delivery of Protein- and Energy-enforced Meals for Older Patients by the Use of ICT-technology
Brief Title: Food'to'Go - a Feasibility Study of Post-discharge Meals for Older Patients by the Use of ICT-technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Tachista (Unknown)
Responsible Party: Principal Investigator, Tove Lindhardt Damsgaard, Senior researcher, Herlev Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-O-FNG-2014-1
Record Dates: First submitted 2014-08-20; First posted 2014-10-20 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Malnutrition
Keywords: Pilot study; Frail elderly; Malnutrition; Functionality; Life quality; Health care technology
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controle Group (No Intervention): Patients in the control group are undergoing the same measurements and records before discharge, and at six and twelve weeks, as the intervention group. The control group receives no special treatment or care after discharge.
- App for food delivery (Other): Intervention: Tablet Computer
  Patients in the intervention group receives a tablet upon discharge from the hospital. The tablet contains an app, which the patients in the intervention group can use for ordering meals for delivery from the kitchen at the hospital three times a week. The app also ask the patients to register their own dietary intake, and give them feedback on their daily energy and protein intake.
  Baseline measurements and records are taken at prior to discharge from the hospital, and after six and twelve weeks.
  Interventions: Device: Tablet computer

INTERVENTIONS:
Device: Tablet computer — Patients receive a tablet computer upon discharge. The tablet can be used for ordering food for delivery three times a week from the hospital kitchen.
  Arms: App for food delivery

SUMMARY:
The research and Innovation program Food'n'Go - Empower aims to develop, test and implement a health technology solution for involvement and increased empowerment of elderly patients and their relatives. The focus is on frequent issues for this group of patients, in the first phase focusing on nutrition and physical activity. Later, the solution will include pain management, management of sleep problems, management of medication, prevention of confusion and coordination of the treatment and care course across sectorial borders. The technology is a tablet-computer, operated by the patient by means of a number of app-like software applications.

The program received in the summer of 2013 one of the Capital Region OPI funding for design and development of the prototype, which is now ready and looking very promising. The next step is a pilot feasibility study testing the usability and acceptability as well as effect during hospitalisation and at home after discharge. The present study - Food'to'Go investigates the intervention in the post-discharge period.

Aim The overall aim of Food'n'Go research- an innovation programme is to develop, test and implement innovative information technology solutions to increase participation and empowerment of older patients and their families, in relation to frequent problems during hospitalisation and the time after.

The aim for the substudy Food'to'Go is to test the feasibility and efficacy of ICT-supported energy- and protein-enforced home-delivered main and in-between meals on older patients, discharged from acute hospitalisation in medical wards. Hereunder:

* Test the technology's relevance, suitability, acceptability and ease of use in relation to the target group
* Test the communication loop between patient and kitchen, and relatives external access to the related website

Welfare and health technologies are often directed at solving problems and meeting the needs of society's most vulnerable groups, often not familiar with computers. We will, in addition to developing the technological solution, examine user-related barriers and preferences for health technology and try to find solutions that can increase older people's possibilities for using technology and achieve empowerment. The program incorporates research and innovation in an iterative process where research provides answers and solutions to the issues arising in relation to the development of the technology (innovation) and the use of it.

ELIGIBILITY:
Inclusion Criteria:

* are 65 years or older
* are admitted to department of internal medicine, O
* have a nutritional risc score of 3 or more
* are discharged to own home
* are able to participate in the project for 12 weeks
* are able to read, write and understand Danish
* live within a radius of 20 km radius from Herlev Hospital

Exclusion Criteria:

* have food allergies or intolerance
* are vegetarians
* are terminally ill
* are included in the RiSK project
* are unable to communicate and co-operate on the use of the tablet computer

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The technology acceptability and ease of use in relation to the target group | 12 weeks
  Method: Registration of how many participants used the technology, as well as registration of the number of problems caused by the technology not working or the participants in-ability to use it.
  Interviews with patients

SECONDARY OUTCOMES:
Test of the communication loop between patient and kitchen | 12 weeks
  Registration of the number of problems caused by lack of communication between devices, or between staff and participants.
Nutritional status | 12 weeks
  BMI and weight
Functional levet | 12 weeks
  Hand-grip strength and chair-stand-test

CONTACTS AND LOCATIONS:
Overall Officials: Tove L Damsgaard, Dr.Med.Sc., Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

REFERENCES:
- See also: Capital region of Denmark's introduction to the project behind the study — http://www.regionh.dk/english/menu/Research+and+Innovation/Innovation/Examples_of_innovation/Food+n+go.htm